CLINICAL TRIAL: NCT03214185
Title: Effects of Preimplantation Genetic Screening 2.0 on the Clinical Outcomes of Assisted Reproductive Treatment in Patients With Recurrent Pregnancy Loss : A Multi-center-based Prospective Randomized Clinical Trial
Brief Title: Effects of PGS2.0 in Patients With Unexplained RPL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Collaborators: The International Peace Maternity & Child Health Hospital of China welfare institute (Unknown); RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JIAI E2017-15
Record Dates: First submitted 2017-07-09; First posted 2017-07-11 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2017-07

CONDITIONS: Recurrent Pregnancy Loss; Infertility, Female
Keywords: unexplained recurrent pregnancy loss; infertility, female; preimplantation genetic screening; in vitro fertilization; intracytoplasmic sperm injection
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With PGS 2.0 (Experimental): Patients will undergo IVF/ICSI procedure, and experience oocyte aspiration, fertilization,blastocyst formation,conventional embryo morphology evaluation and trophectoderm biopsy before blastocyst cryopreservation. Preimplantation genetic screening (PGS) will be performed to select euploid embryo. The patients will go through up to three times of frozen-thawed transfers of euploid blastocysts until ongoing pregnancy or live birth is acquired. Only one euploid blastocyst will be transferred at a time.
  Interventions: Procedure: IVF/ICSI; Genetic: PGS 2.0
- Without PGS 2.0 (Active Comparator): Patients will undergo IVF/ICSI procedure, and experience oocyte aspiration, fertilization,blastocyst formation,and conventional embryo morphology evaluation before blastocyst cryopreservation. The patients will go through up to three times of frozen-thawed transfers of good quality blastocysts until ongoing pregnancy or live birth is acquired. Only one good quality blastocyst will be transferred at a time.
  Interventions: Procedure: IVF/ICSI; Other: Conventional embryo morphology evaluation

INTERVENTIONS:
Procedure: IVF/ICSI — in vitro fertilization or intracytoplasmatic sperm injection
Genetic: PGS 2.0 — Blastocysts are selected by PGS 2.0(NGS based) and only euploid embryos will be transferred.
  Arms: With PGS 2.0
Other: Conventional embryo morphology evaluation — Blastocysts are selected by morphology criteria and only good-scored embryo will be transferred.
  Arms: Without PGS 2.0

SUMMARY:
50%-60% of the known causes of recurrent pregnancy loss(RPL) are associated with embryonic aneuploidy, such that preimplantation genetic screening (PGS) on embryos acquired by assisted reproductive treatment should improve the rate of pregnancy and live birth in those patients. In dispute though the clinical application of PGS has been, a series of studies show that the new generation of PGS(PGS 2.0), based on blastocyst biopsy followed by whole genome analysis, has significantly improved the clinical outcome of IVF treatment. At present, there is still a need for the evidence of the use of PGS 2.0 in RPL patients, who may benefit from this emerging technology considering the prevalence of genetic abnormalities and the number of transferable embryos in this population.

An earlier single center RCT conducted by our IVF center displayed higher implantation rate, clinical pregnancy rate and ongoing pregnancy rate calculated by per embryo transfer(ET) cycle in IVF/ICSI+PGS group compared with IVF/ICSI group.

This multi-center prospective randomized clinical trial is to provide more data to determine whether the clinical outcomes are significantly improved per treatment cycle such that provide evidence for the application of PGS in RPL patients. Besides, risk factors of PGS outcome are to be analyzed from multi-center data to build a model for prediction of the possible outcomes of PGS and direction of the clinical choice.

ELIGIBILITY:
Inclusion criteria:

1. The couple has experienced two or more failed pregnancies (according to ASRM definition).
2. The karyotypes of both husband and wife are normal (polymorphic chromosomes are considered normal either).

3. Women ages ≥20 and <38 years old.

Exclusion criteria:

1. the wife has history of the following diseases: a, the history of thyroid disease; b, the history of adrenal diseases; c, the history of sexually transmitted diseases; d, the history of hereditary diseases; e, the history of mental and psychological disorders.
2. the wife has the following uterine abnormalities: a, uterine malformations (uterus unicorns and duplex uterus), untreated septate uterus, adenomyoma, submucous uterine fibroids, endometrial polyps, or intrauterine adhesions (including the history of intrauterine adhesions).
3. the wife has a medical condition that contraindicate ART or pregnancy, including poorly controlled type I or type II diabetes; undiagnosed liver and renal disease or liver and renal insufficiency (based on blood test); deep vein thrombosis; pulmonary embolism; history of cerebrovascular accident; uncontrolled hypertension; cardiac disease; carcinoma; severe anemia; suspicious or undiagnosed vaginal bleeding.

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 710 (Estimated)
Dates: Start 2018-02-06 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Live birth rate per initiated cycle | up to 42 days of a live birth
  live birth rate of a baby per oocyte retrieval cycle initiated

SECONDARY OUTCOMES:
Embryo implantation | 2 weeks after embryo transfer
  positive serum hCG after 2 weeks of embryo transfer
Clinical pregnancy | 4 weeks after embryo transfer
  the presence of a gestational sac confirmed by transvaginal ultrasound examination
Ongoing pregnancy | 10 weeks after embryo transfer
  the fetal heat beat continued at 10 weeks after embryo transfer
Time to pregnancy | From the day of entering oocyte retrieval cycle to the embryo transfer day of a later assured ongoing pregnancy,which is up to 24 months within the study period.
  From the day of entering oocyte retrieval cycle to the embryo transfer day of a later assured ongoing pregnancy,which is up to 24 months within the study period.If the patient fails to obtain ongoing pregnancy during the study period, this outcome measure will not be recorded.
Pregnancy outcome | up to 42 days of a live birth
  abortion, multiple birth, birth defects, preterm delivery, small for gestational age, still birth

CONTACTS AND LOCATIONS:
Overall Officials: XIAOXI SUN, PHD, Study Chair — Shanghai Ji Ai Genetics & IVF Institute, Obstetrics and Gynecology Hospital, Fudan University
Locations (1):
- Shanghai Ji Ai Genetics & IVF Institute, Obstetrics and Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Practice Committee of the American Society for Reproductive Medicine. Definitions of infertility and recurrent pregnancy loss: a committee opinion. Fertil Steril. 2013 Jan;99(1):63. doi: 10.1016/j.fertnstert.2012.09.023. Epub 2012 Oct 22. PMID 23095139
- [Background] Kolte AM, Bernardi LA, Christiansen OB, Quenby S, Farquharson RG, Goddijn M, Stephenson MD; ESHRE Special Interest Group, Early Pregnancy. Terminology for pregnancy loss prior to viability: a consensus statement from the ESHRE early pregnancy special interest group. Hum Reprod. 2015 Mar;30(3):495-8. doi: 10.1093/humrep/deu299. Epub 2014 Nov 5. PMID 25376455
- [Background] Hodes-Wertz B, Grifo J, Ghadir S, Kaplan B, Laskin CA, Glassner M, Munne S. Idiopathic recurrent miscarriage is caused mostly by aneuploid embryos. Fertil Steril. 2012 Sep;98(3):675-80. doi: 10.1016/j.fertnstert.2012.05.025. Epub 2012 Jun 7. PMID 22683012
- [Background] Scott RT Jr, Upham KM, Forman EJ, Hong KH, Scott KL, Taylor D, Tao X, Treff NR. Blastocyst biopsy with comprehensive chromosome screening and fresh embryo transfer significantly increases in vitro fertilization implantation and delivery rates: a randomized controlled trial. Fertil Steril. 2013 Sep;100(3):697-703. doi: 10.1016/j.fertnstert.2013.04.035. Epub 2013 Jun 1. PMID 23731996
- [Background] Forman EJ, Hong KH, Ferry KM, Tao X, Taylor D, Levy B, Treff NR, Scott RT Jr. In vitro fertilization with single euploid blastocyst transfer: a randomized controlled trial. Fertil Steril. 2013 Jul;100(1):100-7.e1. doi: 10.1016/j.fertnstert.2013.02.056. Epub 2013 Mar 30. PMID 23548942
- [Background] Dahdouh EM, Balayla J, Garcia-Velasco JA. Comprehensive chromosome screening improves embryo selection: a meta-analysis. Fertil Steril. 2015 Dec;104(6):1503-12. doi: 10.1016/j.fertnstert.2015.08.038. Epub 2015 Sep 16. PMID 26385405
- [Background] Dahdouh EM, Balayla J, Garcia-Velasco JA. Impact of blastocyst biopsy and comprehensive chromosome screening technology on preimplantation genetic screening: a systematic review of randomized controlled trials. Reprod Biomed Online. 2015 Mar;30(3):281-9. doi: 10.1016/j.rbmo.2014.11.015. Epub 2014 Dec 11. PMID 25599824
- [Background] Sermon K, Capalbo A, Cohen J, Coonen E, De Rycke M, De Vos A, Delhanty J, Fiorentino F, Gleicher N, Griesinger G, Grifo J, Handyside A, Harper J, Kokkali G, Mastenbroek S, Meldrum D, Meseguer M, Montag M, Munne S, Rienzi L, Rubio C, Scott K, Scott R, Simon C, Swain J, Treff N, Ubaldi F, Vassena R, Vermeesch JR, Verpoest W, Wells D, Geraedts J. The why, the how and the when of PGS 2.0: current practices and expert opinions of fertility specialists, molecular biologists, and embryologists. Mol Hum Reprod. 2016 Aug;22(8):845-57. doi: 10.1093/molehr/gaw034. Epub 2016 Jun 2. PMID 27256483
- [Derived] Lei C, Sui Y, Ye J, Lu Y, Xi J, Sun Y, Jin L, Sun X. Comparison of PGS2.0 versus conventional embryo morphology evaluation for patients with recurrent pregnancy loss: a study protocol for a multicentre randomised trial. BMJ Open. 2020 Oct 7;10(10):e036252. doi: 10.1136/bmjopen-2019-036252. PMID 33033011
- [Derived] Cornelisse S, Zagers M, Kostova E, Fleischer K, van Wely M, Mastenbroek S. Preimplantation genetic testing for aneuploidies (abnormal number of chromosomes) in in vitro fertilisation. Cochrane Database Syst Rev. 2020 Sep 8;9(9):CD005291. doi: 10.1002/14651858.CD005291.pub3. PMID 32898291